CLINICAL TRIAL: NCT03921021
Title: Phase 2 Study of Telomelysin (OBP-301) in Combination With Pembrolizumab in Esophagogastric Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Oncolys BioPharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1807019403
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Esophagogastric Adenocarcinoma
Keywords: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Telomelysin (OBP-301) (Experimental): All patients will receive Telomelysin (OBP-301) at 2x10^12 viral particles (VP)/ tumor injection administered every two weeks x 4 injections as well as standard dose pembrolizumab 200 mg IV every 3 weeks. The tumor will be injected with OBP-301 four times (d1, d15, d29, d43). The preference is to inject the primary tumor endoscopically. Metastatic lesions may be injected on a case-by-case basis after discussion with the PI (Shah).
  Interventions: Drug: Telomelysin

INTERVENTIONS:
Drug: Telomelysin — OBP-301, the investigational product (IP) is formulated in 20 mM Tris pH 8.0, 25 mM NaCl with 2.5% glycerin, USP by volume. OBP-301 will be injected into the target tumor lesions.
  Other Names: OBP-301

SUMMARY:
This is a phase II study of OBP-301 with pembrolizumab in advanced gastric and gastroesophageal junction adenocarcinoma that has progressed on at least 2 lines of prior therapy for advanced disease.

DETAILED DESCRIPTION:
This is a phase II study of OBP-301 with pembrolizumab in advanced gastric and gastroesophageal junction adenocarcinoma that has progressed on at least 2 lines of prior therapy for advanced disease. Pembrolizumab has recently received FDA approval for PD-L1 positive gastric and GEJ adenocarcinoma based on the Keynote-059 study. The efficacy of pembrolizumab monotherapy is modest in PD-L1 positive patients (defined as a combined positive score, CPS, of > 1), with only a ~15% overall response rate. This study will examine the addition of the oncolytic virus, OBP-301, administered prior to pembrolizumab in this patient population. Patients will be enrolled in a two-stage design, with 18 patients in the first stage. All patients will receive OBP-301 at 2x1012 viral particles (VP)/ tumor injection administered every two weeks x 4 injections as well as standard dose pembrolizumab 200 mg IV every 3 weeks. The tumor will be injected with OBP-301 four times (d1, d15, d29, d43). The preference is to inject the primary tumor endoscopically. Metastatic lesions may be injected on a case-by-case basis after discussion with the PI (Shah). All patients treated with OBP-301 will be eligible for the safety cohort.

Primary Endpoints:

* To examine the efficacy of OBP-301 with pembrolizumab in PD-L1 positive advanced gastric and gastroesophageal junction adenocarcinoma in the 3rd or 4th line setting, as assessed by the RECIST response rate.
* To examine the safety of multiple OBP-301 intratumoral injections in combination with pembrolizumab in advanced gastroesophageal adenocarcinoma.

Secondary Endpoint:

• To examine other measures of efficacy of the combination of OBP-301 with pembrolizumab in advanced gastric and esophageal adenocarcinoma including the disease control rate, duration of response, overall survival and progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be >18 years of age on the day of signing the informed consent.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Have histologically or cytologically confirmed advanced or metastatic gastroesophageal adenocarcinoma, at least 1 cm in size and amenable to intratumoral injection.
* Patient must have received at least 2 line of systemic therapy for advanced disease.
* Tumor must be PD-L1 positive, as defined by a combined positive score (CPS).
* Have one or more measurable lesions based on iRECIST.
* Be willing to provide tissue; newly obtained biopsy specimens or formalin-fixed, paraffin-embedded (FFPE) block specimens.
* Female subjects of childbearing potential have a negative urine or serum pregnancy test within 7 days prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. If a serum pregnancy test is required it can be performed on the same day as the urine pregnancy test. The serum pregnancy test must also be completed 7 days prior to enrollment. And male / female subjects of childbearing potential must agree to use an adequate method of contraception starting with signing the informed consent through 120 days after the last dose of study medication.
* Demonstrated adequate organ function as defined in following criteria. All screening labs should be performed within 14 days of enrollment. Note: Subject must not have taken transfusion, hematopoietic agent; granulocyte-colony stimulating factor (GCSF) etc., and/or oxygen supplementation within 7 days before the screening labs.
* Absolute neutrophil count (ANC)>1,000 /mm3
* Platelets>100,000 /mm3
* Hemoglobin>8.0 g/dL
* Serum total bilirubin<2.0 mg/dL
* Aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT)< 3x Upper limit of normal (ULN). For subjects with liver metastases< 5x ULN.
* Serum creatinine< 2.0 mg/dL; or if serum creatinine > 2.0 mg/dL, measured or calculated creatinine/clearance >45 mL/min (Cockcroft-Gault formula).
* Life expectancy of ≥ 4 months from the first OBP-301 treatment.
* Understand the study requirements and the treatment procedures, and is willing to comply with all specified follow-up evaluations, and provides written informed consent before any study-specific tests or procedures are performed.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks of study Day 1.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (greater than equivalent of prednisone 20 mg/day) or any other form of immune-suppressive therapy within 7 days prior to study Day 1.
* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has had prior anti-cancer monoclonal antibody chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1, who has not recovered from adverse events due to a previously administered agent.
* Has a known additional malignancy within 3 years of first injection of OBP-301 that is progressing or requires active treatment, with the exception of prostate cancer controlled with androgen deprivation therapy.
* Has received a live vaccine within 30 days of planned start of study therapy.
* Patients known to have acute or chronic active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
* Has any evidence of active, non-infectious pneumonitis or interstitial lung disease requiring steroids.
* Has an active infection requiring systemic therapy within 2 weeks of Day 1.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Previous severe hypersensitivity to another monoclonal antibody
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled diabetes, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/psychological incompetence, whereby in the opinion of the Investigator the patient is assessed as being unable to provide information, consent, or comply with the study requirements and procedures.
* Patients who are pregnant or breastfeeding, or expecting to conceive or father children within the projected timeframe of the study, starting from the time of the Screening Visit through 4 months (120 days) after the last OBP-301 administration. Females of childbearing potential must have a negative serum or urine pregnancy test at Screening. A female not of childbearing potential is one who has undergone bilateral oophorectomy or who has had no menses for 12 consecutive months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telomelysin (OBP-301)
Started | 17
Completed | 1
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate, as Assessed by Radiographic Imaging
Description: The examination of patients with a partial or complete response is reported as the number of patients who achieved either a complete or partial response (CR + PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Per RECIST v1.1, for target lesions assessed by MRI or CT Chest Abdomen and Pelvis with Contrast, a Complete Response (CR) is the disappearance of all target lesions, and a Partial Response (PR) is a ≥30% decrease in the sum of the longest diameter of target lesions. Overall Response (OR) is defined as the sum of CR and PR.
Time Frame: 1 year
Population: 16 out of 17 enrolled participants were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 16
Participants | 3

2. Secondary Outcome: Disease Control Rate, as Assessed by Radiographic Imaging
Description: Examination of subjects with stable disease, a partial response, or complete response reported as the number of participants who maintained stable disease, partial response, or complete response as per iRECIST through 1 year (SD + PR + CR). The examination of patients with a partial or complete response is reported as the number of patients who achieved either a complete or partial response (CR + PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Per RECIST v1.1, for target lesions assessed by MRI or CT Chest Abdomen and Pelvis with Contrast, a Complete Response (CR) is the disappearance of all target lesions, and a Partial Response (PR) is a ≥30% decrease in the sum of the longest diameter of target lesions. Overall Response (OR) is defined as the sum of CR and PR.
Time Frame: 1 year
Population: 16 out of 17 patients enrolled were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 16
Participants | 4

3. Secondary Outcome: Duration of Response, as Assessed by Radiographic Imaging
Description: Defined as the duration that subjects who have responded to combination therapy remain without disease progression. The examination of patients with a partial or complete response is reported as the number of patients who achieved either a complete or partial response (CR + PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Per RECIST v1.1, for target lesions assessed by MRI or CT Chest Abdomen and Pelvis with Contrast, a Complete Response (CR) is the disappearance of all target lesions, and a Partial Response (PR) is a ≥30% decrease in the sum of the longest diameter of target lesions. Overall Response (OR) is defined as the sum of CR and PR.
Time Frame: 2.5 years
Population: 3 out of 17 enrolled patients were evaluable for duration of response.
Measure: Median (Full Range); unit: days
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 3
days | 498 [461 to 758]

4. Secondary Outcome: Overall Survival Rate, as Assessed by Survival
Description: Defined as the number of participants who survived until 1 year from enrollment
Time Frame: 1 year
Population: 14 out of 17 enrolled participants were evaluable for survival at 1 year from registration.
Measure: Count of Participants; unit: Participants
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 14
Participants | 3

5. Secondary Outcome: Progression Free Survival Rate, as Assessed by Radiographic Imaging and Survival.
Description: The number of participants who did not progress as determined by iRECIST, or die by 1 year. The examination of patients with a partial or complete response is reported as the number of patients who achieved either a complete or partial response (CR + PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Per RECIST v1.1, for target lesions assessed by MRI or CT Chest Abdomen and Pelvis with Contrast, a Complete Response (CR) is the disappearance of all target lesions, and a Partial Response (PR) is a ≥30% decrease in the sum of the longest diameter of target lesions. Overall Response (OR) is defined as the sum of CR and PR.
Time Frame: 1 year
Population: 16 out of 17 participants enrolled were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Telomelysin (OBP-301)
Number analyzed (Participants) | 16
Participants | 3

6. Other Pre Specified Outcome: Change From Baseline in Tumor-immune Microenvironment, as Measured by Bulk RNA Sequencing and Single-cell RNA Sequencing.
Description: In this aim we will summarize the results from all patient data to assess what are the consistent changes observed in cellular composition in response to immunotherapy and we will investigate how these changes impact response to treatment.
Time Frame: Baseline, 2 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change From Baseline in T-cell Response, as Measured by TCR-sequencing of Tumor Biopsies
Description: This project will be focused on analyzing the immune landscape of individual tumors from tumor biopsies taken at baseline and on therapy. We will analyze changes associated with relapse and differences between refractory and sensitive patients. Our proposed analysis will take as input somatic mutations, raw WES reads, and raw RNA-Seq reads
Time Frame: Baseline, 2 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change From Baseline in Immune Infiltrate by Multi-parameter Flow-cytometry
Description: This powerful approach will be utilized to characterize tumor immune cell infiltrates at baseline, following the induction of combination therapy and at the time of resection. This will be one of the first longitudinal analyses of tumor immune cell infiltrates by multi-parameter flow cytometry following immunotherapy.
Time Frame: Baseline, 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected until 30 days following last dose of study drug for a maximum of approximately 2 years.
Arm/Group | Telomelysin (OBP-301)
All-Cause Mortality (participants affected / at risk) | 13/17
Serious Adverse Events (participants affected / at risk) | 15/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telomelysin (OBP-301) (N=17)
Other: Gastrointestinal Bleed (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Other: Muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Other: Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Sepsis (Infections and infestations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Pericardial Tamponade (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Fever (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telomelysin (OBP-301) (N=17)
Anemia (Blood and lymphatic system disorders) | 3
Acute coronary syndrome (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Other - Ear and labyrinth disorders (Decreased hearing) (Ear and labyrinth disorders) | 1
Dry Eye (Eye disorders) | 1
Others - Eye disorders (Intermittent Vision fogginess and Left-sided eye lid lag) (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Esophagitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 6
Other - Gastrointestinal disorder (Gastrointestinal bleed) (Gastrointestinal disorders) | 2
Other - Gastrointestinal disorder (Dark stool) (Gastrointestinal disorders) | 1
Other - Gastrointestinal disorder (Epigastric pain and Abdominal Mass) (Gastrointestinal disorders) | 1
Other - Gastrointestinal disorder (Small bowel obstruction) (Gastrointestinal disorders) | 1
Other - Gastrointestinal disorder (Dry heaving) (Gastrointestinal disorders) | 1
Other - Gastrointestinal disorder (Abdominal tenderness) (Gastrointestinal disorders) | 1
Other - Gastrointestinal disorder (Belching) (Gastrointestinal disorders) | 1
Other - Gastrointestinal disorder (Melena) (Gastrointestinal disorders) | 1
Other - Gastrointestinal disorder (Balance Issues) (Gastrointestinal disorders) | 1
Chills (General disorders) | 4
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 7
Fever (General disorders) | 5
Flu like symptoms (General disorders) | 1
Other (Delayed Speech and Ill-appearing ) (General disorders) | 1
Other (Cold Sore, Edema and Localized pain near injection site) (General disorders) | 1
Other (lightheadedness) (General disorders) | 1
Other (Cervical Adenopathy) (Immune system disorders) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Weight loss (Investigations) | 3
Other (Blood urea nitrogen increased) (Investigations) | 1
Other (Hyponatremia) (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 3
Other (Hyponatremia) (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Other (Pain to left ribs) (Musculoskeletal and connective tissue disorders) | 1
Other (Body Aches) (Musculoskeletal and connective tissue disorders) | 1
Other (Left flank pain) (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Other (Cranial face deficit and Facial asymmetry) (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 2
Hallucinations (Psychiatric disorders) | 1
Other (Nervousness) (Psychiatric disorders) | 1
Other (Slow behavior and Distress) (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Other (Rectal bleeding) (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Other- Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Other (Pallor) (Skin and subcutaneous tissue disorders) | 1
Other (Small pustule on scrotum) (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT03921021/Prot_SAP_000.pdf